CLINICAL TRIAL: NCT01780792
Title: Examining the Effects of Dance, Dance Revolution on Mobility, Brain Plasticity and Cognition in Individuals With Multiple Sclerosis
Brief Title: Examining the Effects of Video-game Exercise on Mobility and Brain Plasticity in Individuals With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ruchika Prakash, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011H0048
Record Dates: First submitted 2012-11-07; First posted 2013-01-31 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; mobility; cognition; neuroplasticity; videogame play
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dance Dance Revolution game play (Experimental): Dance Dance Revolution video game play
  Interventions: Other: Dance Dance Revolution video game play
- control (No Intervention): individuals continue usual care for 8 weeks

INTERVENTIONS:
Other: Dance Dance Revolution video game play — Individuals play dance dance revolution 3 times a week for 8 weeks
  Arms: Dance Dance Revolution game play

SUMMARY:
Dance Dance Revolution (DDR) may offer an innovative and highly effective format for delivering exercise programs to people with multiple sclerosis (MS). It is a fun, engaging and interactive video game that requires players to move their feet to targets while matching the rhythm of a song. In addition, DDR, involving both aerobic exercise and cognitive training, is an ideal intervention for improving cognitive functioning in those with MS. The purpose of this pilot study is to examine the use of DDR as a novel and highly specific exercise intervention to improve mobility and cognition among individuals with MS.

DETAILED DESCRIPTION:
Dance Dance Revolution (DDR) may offer an innovative and highly effective format for delivering exercise programs to people with MS. It is a fun, engaging and interactive video game that requires players to move their feet to targets while matching the rhythm of a song. In addition, DDR, involving both aerobic exercise and cognitive training, is an ideal intervention for improving cognitive functioning in those with MS. The purpose of this pilot study is to examine the use of DDR as a novel and highly specific exercise intervention to improve mobility and cognition among individuals with MS. We will be guided by the following three specific aims and hypotheses:

Specific Aim 1: Determine if an eight-week exercise program administered using DDR improves dynamic balance in people with MS relative to a wait-list control group.

Hypothesis 1: Dynamic balance as measured by the Berg Balance Scale will be more improved with the DDR intervention than the wait-list control group.

Specific Aim 2: Determine if the DDR intervention, combining fitness and cognitive training, over the course of an eight-week intervention, will have a more positive effect on domains of processing speed and executive control, than a wait-list control group.

Hypothesis 2: The DDR group relative to the wait-list control group, will show significant improvement in cognitive functioning as assessed by the Paced Auditory Serial Addition Test (PASAT), a measure of processing speed, and executive functioning. Specifically, we hypothesize that given severe deficits in processing speed and executive control, participation in a DDR intervention, will result in a significant improvement on the PASAT, a widely used measure to assess cognitive functioning in patients with MS.

Specific Aim 3: We will also examine whether improvements in cognitive processes engendered by DDR on the PASAT will be supported by changes in underlying neural circuits, as inferred from patterns of event-related functional magnetic resonance imaging (fMRI) activation obtained in a 3 Tesla scanner.

Hypothesis 3: Improvements in cognition as indexed by higher accuracy scores and faster reaction time on the PASAT, will be accompanied by a change in the recruitment of underlying neural processes as inferred from functional magnetic resonance imaging. MS participants in the DDR group will show an increase in recruitment of the attentional network, and more specifically the prefrontal and parietal cortices, cortical regions responsible for successful performance on the PASAT task.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Score of < 5 and a diagnosis of relapsing-remitting multiple sclerosis

Exclusion Criteria:

* other neurological or orthopedic diagnosis that limits ambulation, age 30-59

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | after 8 weeks
  The Berg Balance scale consists of 14 functional activities that test static and dynamic balance. Each item is scored on a scale of 0-4 with higher scores indicating better balance
PASAT | after 8 weeks
  The PASAT is a measure of sustained attention, working memory and information processing speed.

SECONDARY OUTCOMES:
4 square step test | after 8 weeks
  requires a person to step rapidly in a multi-directional pattern over a cane. It predicts fallers
The Activities Specific Balance Confidence Scale | after 8 weeks
  Measures fear of falling. Subjects rate their balance confidence on 10 items.
GAITRite | after 8 weeks
  individuals walk on a computerized carpet that records spatiotemporal aspects of gait such as velocity and stride length.
6 minute walk test | Immediately prior to starting the intervention/control period,, after 8 week intervention/control period and then at an 8 week follow up
  subjects walk for 6 minutes and distance walked is measured
physical activity | after 8 weeks
  subjects wear an accelerometer for 5 days which records how active they are.
multiple sclerosis quality of life inventory | after 8 weeks
  the MS quality of life inventory is filled out to measure the impact of MS on the individuals quality of life.
fMRI | after 8 weeks
  individuals will go into an MRI and undergo neuropsychological and motor testing to examine for neuroplasticity

CONTACTS AND LOCATIONS:
Overall Officials: Deb Kegelmeyer, DPT, MS, Principal Investigator — Ohio State University; Ruchika Prakash, PhD, Principal Investigator — Ohio State University; Anne Kloos, PT, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Atwell Hall, Columbus, Ohio, United States